CLINICAL TRIAL: NCT02199158
Title: Short-term Outcomes of Iridoplasty for Persistent Angle Closure Despite Patent Iridotomies An Anterior Segment Optical Coherence Tomography Study
Brief Title: Short-term Outcomes of Iridoplasty for Persistent Angle Closure Despite Patent Iridotomies
Acronym: ALPIECA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: iridoplastiaeca
Record Dates: First submitted 2014-07-14; First posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Angle Closure Glaucoma; Glaucoma
Keywords: iridoplasty; angle; glaucoma; anterior chamber; laser treatment
MeSH Terms: conditions — Glaucoma, Angle-Closure; Glaucoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Argon Laser Peripheral Iridoplasty (Experimental): ALPI was applied with a VISULAS diode laser of 532 nm (Carl Zeiss Meditec, Dublin, CA) by the same ophthalmologist (JML). Twenty to 40 spots of 400 mW power with 500 microns of size and duration of 500 ms were applied. Power was modified arbitrarily until an effective iris contraction was obtained. It was considered an effective contraction as that which causes a concentric movement around the laser spot, with minimal iris pigmentation and immediate angle opening observed through the lens mirrors using a Goldmann lens. Power was lowered if there was any bursting sound perceived, pigment dispersion, air bubbles or considerable pain.
  Interventions: Procedure: Argon Laser Peripheral Iridoplasty

INTERVENTIONS:
Procedure: Argon Laser Peripheral Iridoplasty — ALPI was applied with a VISULAS diode laser of 532 nm (Carl Zeiss Meditec, Dublin, CA) by the same ophthalmologist (JML). Twenty to 40 spots of 400 mW power with 500 microns of size and duration of 500 ms were applied. Power was modified arbitrarily until an effective iris contraction was obtained. It was considered an effective contraction as that which causes a concentric movement around the laser spot, with minimal iris pigmentation and immediate angle opening observed through the lens mirrors using a Goldmann lens. Power was lowered if there was any bursting sound perceived, pigment dispersion, air bubbles or considerable pain.
  Other Names: ALPI; Iridoplasty

SUMMARY:
Purpose:

To evaluate short-term angle opening after argon peripheral iridoplasty using AS-OCT and to report its complications at 1-week and 1-month follow up in patients that did not achieve a satisfactory clinical angle opening despite patent laser peripheral iridotomy.

Design:

Prospective, Interventional case series

Subjects:

Patients with an occludable angle in more than two quadrants in dark room indentation gonioscopy and patent iridotomies of at least 2 weeks, with assessment of persistent angle closure aetiology by ultrabiomicroscopy and A-scan ultrasound are included.

Patients will undergo complete examination and AS-OCT before ALPI, one week and one month after it. We analyzed the images in a masked manner and took the angle measurements (AOD500, AOD 750, TISA500, TISA750, ARA500, ARA 750, Lens vault) at 0° and 180° as the main outcome measure to determine effectiveness.

DETAILED DESCRIPTION:
Background Argon laser peripheral iridoplasty (ALPI) (Figure 1) is an iris-remodeling procedure that intends to widen the iridocorneal angle through redistribution of peripheral iris tension forces close to the trabeculum.

ALPI is effective in patients with plateau iris syndrome and acute angle closure glaucoma but there is less published about its effectiveness in secondary angle closure. Therefore, we are going to evaluate this procedure in those patients that did not achieve a satisfactory clinical angle opening despite patent laser peripheral iridotomy, as long as there was no contraindication for a new laser procedure and provided that cataract surgery is not viable, as in clear lens or patients not willing to undergo surgery.

To evaluate its effectiveness, we will use a non-invasive non-contact method through anterior segment optical coherence tomography (AS-OCT), which transmits and receives light in an ultrasound-like manner to obtain anterior segment imaging that helps to evaluate the angle more objectively.

Purpose To evaluate short-term angle opening after argon peripheral iridoplasty using AS-OCT and to report its complications at 1-week and 1-month follow up in patients with persistent angle closure despite patent iridotomies.

Study Design Prospective, interventional case series Patients with an occludable angle in more than two quadrants in dark room dynamic gonioscopy and patent iridotomies of at least 2 weeks were included. A supplemental diagnosis regarding the etiology of persistent angle closure by ultrabiomicroscopy and A-scan ultrasound will be obtained. Patients who presented with these criteria to the angle closure clinic at the glaucoma service of our institute (Instituto de Oftalmologia Fundacion Conde de Valenciana IAP, Mexico City) between July and November 2012 were included.

Patients with synechiae of more than one quadrant, advanced glaucomatous damage, prompt cataract surgery plans and those who did not wish to participate were excluded.

After obtaining informed consent, patients underwent biomicroscopy, gonioscopy, visual acuity, intraocular pressure and AS-OCT before ALPI, one week and one month after it. The AS-OCT Visante (Carl Zeiss Meditec, Dublin) took an image of the vertical and horizontal meridians at the same room illumination of 14 lux measured with a luxometer mobile application (Apple Inc., Application Manufactory available at the AppStore by June 2012).

Images were analyzed in a masked manner marking scleral spurs and angle recess at 0° and 180° of the horizontal image.

ALPI was applied with a VISULAS diode laser of 532 nm (Carl Zeiss Meditec, Dublin, CA) by the same ophthalmologist (JML). Twenty to 40 spots of 400 mW power with 500 microns of size and duration of 500 ms were applied. Power was modified arbitrarily until an effective iris contraction was obtained. It was considered an effective contraction as that which causes a concentric movement around the laser spot, with minimal iris pigmentation and immediate angle opening observed through the lens mirrors using a Goldmann lens. Power was lowered if there was any bursting sound perceived, pigment dispersion, air bubbles or considerable pain. Pilocarpine was not applied before the procedure in all cases because some eyes had angle closure secondary to ciliary block and we considered it could worsen the closure in many cases.

Topical prednisolone acetate was applied every 4 hours for 1 week and brimonidine tartrate every 12 hours for 1 week .

ELIGIBILITY:
Inclusion Criteria:

* Patients with an occludable angle in more than two quadrants in dark room dynamic gonioscopy and patent iridotomies of at least 2 weeks were included
* A supplemental diagnosis regarding the etiology of persistent angle closure by ultrabiomicroscopy and A-scan ultrasound was obtained.

Exclusion Criteria:

* Patients with synechiae of more than one quadrant
* Advanced glaucomatous damage
* Prompt cataract surgery plans and those who did not wish to participate were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Angle Aperture | 1 month
  Angle opening measured by anterior segment optical coherence tomography

SECONDARY OUTCOMES:
Complications | 1 month
  complications reported by patient and/or examiner

CONTACTS AND LOCATIONS:
Overall Officials: Jorge-Emmanuel Morales-León, MD, Principal Investigator — "Fundación Conde de Valenciana" Ophthalmology Institute
Locations (1):
- "Fundación Conde de Valenciana" Ophthalmology Institute, Mexico City, Obrera, Mexico

REFERENCES:
- [Background] Ritch R, Tham CC, Lam DS. Argon laser peripheral iridoplasty (ALPI): an update. Surv Ophthalmol. 2007 May-Jun;52(3):279-88. doi: 10.1016/j.survophthal.2007.02.006. PMID 17472803
- [Background] Ritch R, Tham CC, Lam DS. Long-term success of argon laser peripheral iridoplasty in the management of plateau iris syndrome. Ophthalmology. 2004 Jan;111(1):104-8. doi: 10.1016/j.ophtha.2003.05.001. PMID 14711720
- [Background] Fu J, Qing GP, Wang NL, Wang HZ. Efficacy of laser peripheral iridoplasty and iridotomy on medically refractory patients with acute primary angle closure: a three year outcome. Chin Med J (Engl). 2013 Jan;126(1):41-5. PMID 23286475